CLINICAL TRIAL: NCT01319942
Title: Combined Radiotherapy and Sorafenib in Patients With Hepatoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Shang-Wen Chen, China Medical University Hospital
Other Study IDs: RT-sorafenib
Record Dates: First submitted 2010-07-20; First posted 2011-03-22 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Radiotherapy; Sorafenib; Treatment outcome
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Unresectable hepatoma: Unresectable hepatoma, unsuitable for transarterial embolization or local failure after transarterial embolization
  Interventions: Other: Radiotherapy combined with sorafenib

INTERVENTIONS:
Other: Radiotherapy combined with sorafenib — Radiotherapy: 46 Gy to 60 Gy prescribed to involved hepatic tumor Sorafenib: 2 tablet of sorafenib (200mg) twice daily (totally 800mg per day)
  Other Names: Radiotherapy with sorafenib

SUMMARY:
This study aims to test the efficacy of combined radiotherapy and sorafenib in patients with locally advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a common cause of cancer mortality in Asia. Most patients present with intermediate or advanced disease. Percutaneous ethanol injection, radiofrequency ablation, and transcatheter arterial chemoembolization (TACE) are not considered as a curative treatment and have achieved very limited success in eradicating large HCC. With the development of new radiotherapy (RT) technique, RT can be more safely given to patients with larger tumor burden. Thus, TACE combined with RT has been suggested for treating large HCC. Based on the results of these studies, RT could achieve a tumor response rate of 50 % to 70 %. However, it has not been definitively shown to prolong the overall or disease-free survival due to lack of a phase III clinical trial. In contrast, a retrospective clinical investigation with molecular study suggests that sublethal dose of RT promoted HCC growth outside RT field.

Two phase III trials were shown to be efficacious and well-tolerated in patients with advanced HCC. Median overall survival was significantly 2 to 3 months longer in the sorafenib group than that in the placebo. It is interesting to recognize the combined therapeutic effect of RT with sorafenib. Based on several preclinical experiments, tumor angiogenesis inhibitors seem to be synergistic with irradiation when using before RT, concurrently with RT, or after RT. Thus, we design a single-arm phase II clinical trial to investigate the efficacy of combined RT with sorafenib.

The eligibility criteria are patients with unresectable HCC; good performance status; no prior radiotherapy for the liver; clinical measurable tumor; good liver function and good compliance. After entering this study, the testee will receive RT to hepatic tumor with concurrently sorafenib with a dose of 400 mg twice daily. Hepatic RT will be performed with a daily fraction size of 2.0 to 2.5 Gy to a total dose of 46 Gy to 60 Gy. After RT, maintenance sorafenib with a dose of 400 mg twice daily will be ongoing. Sorafenib will be continued until the occurrence of clinical or radiologic progression, or the occurrence of either unacceptable adverse events or death. Minimum maintenance duration of 6 months is recommended, but not mandatory. The primary end points are response rate and toxicities profile. The secondary endpoints are time to radiological progression interval (TRPI), overall survival, and quality of life assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable hepatoma with transarterial embolization (TAE) failure or who are not suitable for TAE.
2. Age: 20 ~ 69 years.
3. ECOG 0 or 1.
4. Life expectancy of at least 12 weeks.
5. Child-Pugh A or B (preferentially score ≦ 7).
6. Cancer of the Liver Italian Program (CLIP) score ≦ 3.
7. Pretreatment liver function test and renal function test:

   * Total bilirubin < 1.5 times the upper limit of normal (ULN)≦ 3.0(ULN)in patients treated by biliary drainage for obstructive jaundice.
   * GOP/GPT ≦ 5 X of upper limit of normal range.
   * Alkaline phosphatase ≦ 4X of upper limit of normal range.
   * Prothrombin time/partial prothrombin time < 1.5 X of ULN.
   * Serum Creatinine ≦ 1.0 x ULN.
8. Pretreatment blood count:

   * Hemoglobulin ≧ 9 g/dl.
   * Absolute neutrophil count ≧ 1500/mm3.
   * Platelet count ≧ 100,000/mm3.
9. Subjects with at least one uni-dimensional or bi-dimensional measurable lesion. Lesion must be measured by CT scan or MRI.
10. Patients must fully recover from prior therapy that given > 4 weeks before enrolment.11. Signed informed consent must be obtained prior to any study related procedures.

Exclusion Criteria:

1. Child-Pugh C
2. CLIP score ≧ 4
3. Patients with evidence of extrahepatic or metastatic disease
4. Patients with evidence of massive ascites
5. Patients receiving previous irradiation to liver
6. Patients with previous use of Thalidomide less than 6 months from entering of the study
7. History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrythmias requiring anti-arrythmic therapy (beta blockers or digoxin are permitted)
8. Active clinically serious infections ( > grade 2 CTC version 2)
9. Patients undergoing renal dialysis
10. Patients with evidence or history of bleeding diathesis
11. Prior treatment with EGFR TKIs or VEGFR TKIs
12. Hypertension uncontrolled by medical therapy
13. Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry. Also the patient must not be undergoing acute steroid therapy or taper.
14. Chemotherapy or immunotherapy or other systemic anti-cancer therapy within 4 weeks (6 weeks for nitrosoureas, mitomycin and suramin)
15. Major surgery within 4 weeks of start of study
16. Concomitant treatment with strong CYP3A4 inducers or inhibitors
17. Investigational drug therapy outside of this trial during or within 4 weeks of study entry
18. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
19. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation, including the 30 days period after last study drug dosing.
20. Pregnant or breast-feeding patients
21. Known or suspected allergy to the investigational agent or any agent given in association with this trial
22. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry
23. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
24. Patients with seizure disorder requiring medication
25. History of organ allograft
26. Use of biologic response modifiers, such as G-CSF, within 3 week of study entry
27. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
28. Autologous bone marrow transplant or stem cell rescue within 4 months of study
29. Patients unable to swallow oral medications

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 patients withunresectable hepatoma
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Response rate | 1-month and 6-month response rate
  1. Response rate at 1-month and 6-month after radiotherapy.
  2. Toxicities profile of combinede treatment

SECONDARY OUTCOMES:
Time-to radiological progression interval | 2-years
  1. Time-to radiological progression interval
  2. 2-year overall survival
  3. 2-year progression-free survival
  4. Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Wen Chen, MD, Principal Investigator — Department of Radiation Oncology, China Medical University Hospital
Locations (2):
- Taiwan (2):
  - Chi-Mei Hospital, Tainan, Taiwan
  - Taipei Medical University Hospital, Taipei, Taiwan